CLINICAL TRIAL: NCT02753699
Title: A Multi-centre Long Term Follow-up Study to Assess the Durability of Sustained Virologic Response in Alisporivir-treated Chronic Hepatitis C Patients
Brief Title: Long Term Follow-up Study to Assess Durability of Sustained Virologic Response in Alisporivir-treated Hepatitis C Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Debiopharm International SA (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: CDEB025A2312; 2011-006131-38 (EudraCT Number)
Record Dates: First submitted 2016-03-16; First posted 2016-04-28 (Estimated); Results first posted 2016-08-26 (Estimated); Last update posted 2016-08-26 (Estimated); Status verified 2016-07

CONDITIONS: Hepatitis C
Keywords: Chronic hepatitis C
MeSH Terms: conditions — Hepatitis C; Hepatitis C, Chronic | interventions — alisporivir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- From Study 2210 (Experimental): All participants enrolled from CDEB025A2210 (n=164) who had been treated with alisporivir during the feeder study. There was no investigational treatment given to participants while enrolled in this follow-up study.
  Interventions: Drug: Alisporivir
- From Study 2301 (Experimental): All participants enrolled from CDEB025A2301 (n=397) who had been treated with alisporivir during the feeder study. There was no investigational treatment given to participants while enrolled in this follow-up study.
  Interventions: Drug: Alisporivir
- From Study 2211 (Experimental): All participants enrolled from CDEB025A2211 (n=162) who had been treated with alisporivir during the feeder study. There was no investigational treatment given to participants while enrolled in this follow-up study.
  Interventions: Drug: Alisporivir

INTERVENTIONS:
Drug: Alisporivir — Intervention of interest; follow-up after ALV-active study
  Other Names: DEB025; Debio 025; ALV

SUMMARY:
The purpose of this study is to follow-up with participants from feeder studies who achieved sustained virologic response (SVR) over 24 hours posttreatment (SVR24), to assess durability of SVR, and to assess the changes in liver disease, development of hepatocellular carcinoma and post-treatment safety over time.

Participants enter this study from feeder studies CDEB025A2210 (NCT01183169), CDEB025A2301 (NCT01318694), and CDEB025A2211 (NCT01215643). They return to the site for up to 48 weeks with a maximum of 3 visits. No treatment is involved.

ELIGIBILITY:
Inclusion Criteria:

1. Provides written informed consent before any assessment is performed
2. Is male or female aged ≥18
3. Has previously completed a Novartis-sponsored hepatitis C study and received alisporivir
4. Has achieved SVR24
5. Is able to comply with the visit schedule

Exclusion Criteria:

1. Use of any investigational drugs within 5 half-lives of enrollment, or within 30 days of that medication, whichever is longer.
2. Use or planned use to start a new course of hepatitis C therapy.
3. No additional exclusions are to be applied by the Investigator, in order to ensure that the study population is representative of all eligible patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 723 (Actual)
Dates: Start 2011-12; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (103):
- United States (12):
  - Novartis Investigative Site, La Jolla, California
  - Novartis Investigative Site, San Diego, California
  - Novartis Investigative Site, Ventura, California
  - Novartis Investigative Site, Bradenton, Florida
  - Novartis Investigative Site, Honolulu, Hawaii
  - Novartis Investigative Site, Springfield, Illinois
  - Novartis Investigative Site, Indianapolis, Indiana
  - Novartis Investigative Site, Arlington, Texas
  - Novartis Investigative Site, Dallas, Texas
  - Novartis Investigative Site, Houston, Texas
  - Novartis Investigative Site, San Antonio, Texas
  - Novartis Investigative Site, Salt Lake City, Utah
- Novartis Investigative Site, Buenos Aires, Buenos Aires, Argentina
- Australia (5):
  - Novartis Investigative Site, Kingswood, New South Wales
  - Novartis Investigative Site, Kogarah, New South Wales
  - Novartis Investigative Site, Westmead, New South Wales
  - Novartis Investigative Site, Greenslopes, Queensland
  - Novartis Investigative Site, Fitzroy, Victoria
- Novartis Investigative Site, Ghent, Belgium
- Canada (3):
  - Novartis Investigative Site, Calgary, Alberta
  - Novartis Investigative Site, Vancouver, British Columbia
  - Novartis Investigative Site, Torono, Ontario
- France (5):
  - Novartis Investigative Site, Clichy
  - Novartis Investigative Site, Créteil
  - Novartis Investigative Site, Lyon
  - Novartis Investigative Site, Nice
  - Novartis Investigative Site, Paris
- Germany (9):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Cologne
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Freiburg im Breisgau
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Kiel
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, Mainz
- Novartis Investigative Site, Hong Kong, Hong Kong, Hong Kong
- Hungary (6):
  - Novartis Investigative Site, Békéscsaba
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Debrecen
  - Novartis Investigative Site, Kaposvár
  - Novartis Investigative Site, Pécs
  - Novartis Investigative Site, Székesfehérvár
- India (4):
  - Novartis Investigative Site, Hyderabad, Andhra Pradesh
  - Novartis Investigative Site, Mumbai, Maharashtra
  - Novartis Investigative Site, Delhi, National Capital Territory of Delhi
  - Novartis Investigative Site, Ludhiana, Punjab
- Italy (11):
  - Novartis Investigative Site, Bologna, BO
  - Novartis Investigative Site, Brescia, BS
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Rozzano, MI
  - Novartis Investigative Site, Palermo, PA
  - Novartis Investigative Site, Parma, PR
  - Novartis Investigative Site, Pavia, PV
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Torino, TO
  - Novartis Investigative Site, Bologna
  - Novartis Investigative Site, Napoli
- Mexico (2):
  - Novartis Investigative Site, Mexico City, Mexico City
  - Novartis Investigative Site, Monterrey, Nuevo León
- Poland (5):
  - Novartis Investigative Site, Bialystok
  - Novartis Investigative Site, Bydgoszcz
  - Novartis Investigative Site, Lódz
  - Novartis Investigative Site, Warsaw
  - Novartis Investigative Site, Zawiercie
- Romania (3):
  - Novartis Investigative Site, Bucharest
  - Novartis Investigative Site, Craiova
  - Novartis Investigative Site, Iași
- Russia (2):
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Saint Petersburg
- South Korea (7):
  - Novartis Investigative Site, Busan, Busan
  - Novartis Investigative Site, Seongnam-si, Gyeonggi-do
  - Novartis Investigative Site, Yangsan, Gyeongsangnam-do
  - Novartis Investigative Site, Seoul, Korea
  - Novartis Investigative Site, Busan
  - Novartis Investigative Site, Incheon
  - Novartis Investigative Site, Pusan
- Spain (4):
  - Novartis Investigative Site, Seville, Andalusia
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Majadahonda, Madrid
  - Novartis Investigative Site, Valencia, Valencia
- Taiwan (8):
  - Novartis Investigative Site, Chiayi City, Taiwan
  - Novartis Investigative Site, Douliu
  - Novartis Investigative Site, Kaohsiung City
  - Novartis Investigative Site, Keelung
  - Novartis Investigative Site, Linkou District
  - Novartis Investigative Site, Niaosong Township
  - Novartis Investigative Site, Taichung
  - Novartis Investigative Site, Taipei
- Thailand (4):
  - Novartis Investigative Site, Bangkok
  - Novartis Investigative Site, Chiang Mai
  - Novartis Investigative Site, Khon Kaen
  - Novartis Investigative Site, Songkhla
- Turkey (Türkiye) (2):
  - Novartis Investigative Site, Fatih / Istanbul
  - Novartis Investigative Site, Izmir
- United Kingdom (6):
  - Novartis Investigative Site, Birmingham
  - Novartis Investigative Site, Glasgow - Scotland
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Newcastle upon Tyne
  - Novartis Investigative Site, Nottingham
  - Novartis Investigative Site, Plymouth
- Vietnam (2):
  - Novartis Investigative Site, Hanoi
  - Novartis Investigative Site, Ho Chi Minh City

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in 127 centers across 22 countries globally.
Pre-assignment Details: Participants transferring from Study 2211 were allocated to the "From Study 2211 group". These were evaluated as INF-free and Overall subgroups for efficacy analyses.
Groups:
- From Study 2210: All participants enrolled from CDEB025A2210 (n=164) who had been treated with alisporivir during the feeder study.
- From Study 2301: All participants enrolled from CDEB025A2301 (n=397) who had been treated with alisporivir during the feeder study.
- From Study 2211: All participants enrolled from CDEB025A2211 (n=162) who had been treated with alisporivir during the feeder study.
Period: Overall Study
Arm/Group | From Study 2210 | From Study 2301 | From Study 2211
Started | 164 | 397 | 162
Completed | 150 | 354 | 139
Not Completed | 14 | 43 | 23

BASELINE CHARACTERISTICS:
Population: The Safety Set, defined as including all patients who had at least one safety observation (adverse event (AE), vital sign and/or laboratory assessment), unless excluded due to protocol deviations.
Groups:
- Total: Total of all reporting groups
Arm/Group | From Study 2210 | From Study 2301 | From Study 2211 | Total
Number analyzed (Participants) | 164 | 397 | 162 | 723
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.5 (9.89) | 46.4 (11.70) | 43.7 (10.89) | 47.2 (11.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58 | 182 | 61 | 301
  Male | 106 | 215 | 101 | 422

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Maintaining Hepatitis C Virus (HCV) Ribonucleic Acid (RNA) Load Below the Level of Quantification (LOQ) Through Week 48
Time Frame: up to 120 Weeks
Population: Full analysis set (FAS), defined as all participants who enrolled into this study and had at least one HCV RNA assessment, unless excluded due to protocol deviations.
Measure: Number; unit: percentage of participants
Groups:
- From Study 2211 IFN-free: Participants enrolled from CDEB025A2211 (n=54) who had been treated with alisporivir in interferon-free (INF-free) regimens during the feeder study.
- From Study 2211 Overall: All participants enrolled from CDEB025A2211 (n=162) who had been treated with alisporivir during the feeder study.
Arm/Group | From Study 2210 | From Study 2301 | From Study 2211 IFN-free | From Study 2211 Overall
Number analyzed (Participants) | 161 | 383 | 53 | 160
percentage of participants
  Week 1 (n=152,371,53,152) | 96.7 | 99.5 | 100.0 | 100.0
  Week 24 (n=148,346,49,148) | 100.0 | 100.0 | 98.0 | 99.3
  Week 48 (n=146,337,46,140) | 100.0 | 99.7 | 100.0 | 100.0
  Week 96 (n=7,0,36,90) | 100.0 | 0.0 | 100.0 | 100.0
  Week 120 (n=0,0,1,3) | 0.0 | 0.0 | 100.0 | 100.0
  Overall (n=161,383,53,160) | 96.9 | 99.2 | 98.1 | 99.4

2. Secondary Outcome: Percentage of Participants With Normal Alanine-aminotransferase (ALT) Values at Week 48.
Description: Note that the 24-week period between end of feeder study (SVR24) and first visit in this follow-up study is not counted in the 48 weeks, so this timepoint corresponds to 96 weeks (=24+24+48) after the last dose of alisporivir.
Time Frame: at Week 48
Population: Full analysis set. In the categories, n is the number of subjects in FAS in the appropriate study group with normal ALT at visit; for Overall - at all available visits.
Measure: Number; unit: percentage of participants
Arm/Group | From Study 2210 | From Study 2301 | From Study 2211 IFN-free | From Study 2211 Overall
Number analyzed (Participants) | 161 | 383 | 53 | 160
percentage of participants
  Week 1 (n=161,383,50,156) | 88.8 | 94.0 | 96.0 | 95.5
  Week 24 (n=150,360,50,151) | 84.0 | 93.9 | 82.0 | 89.4
  Week 48 (n=152,355,47,141) | 88.2 | 91.5 | 87.2 | 91.5
  Week 96 (n=7,0,36,92) | 85.7 | 0.0 | 94.4 | 93.5
  Week 120 (n=0,0,1,3) | 0.0 | 0.0 | 100.0 | 100.0
  Overall (n=161,383,52,159) | 78.9 | 88.5 | 78.8 | 83.6

ADVERSE EVENTS:
Time Frame: Up to 48 weeks
Description: Non-serious adverse events did not reach the 5% reporting threshold.
Arm/Group | From Study 2210 | From Study 2301 | From Study 2211 IFN-free | From Study 2211 Overall
Serious Adverse Events (participants affected / at risk) | 7/164 | 8/397 | 1/54 | 3/162
Other Adverse Events (participants affected / at risk) | 0/164 | 0/397 | 0/54 | 0/162
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | From Study 2210 (N=164) | From Study 2301 (N=397) | From Study 2211 IFN-free (N=54) | From Study 2211 Overall (N=162)
Hypochromic anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Herpes simplex meningitis (Infections and infestations) | 0 | 1 | 0 | 0
Meningitis viral (Infections and infestations) | 0 | 1 | 0 | 0
Osteomyelitis acute (Infections and infestations) | 0 | 1 | 0 | 0
Otitis media chronic (Infections and infestations) | 0 | 1 | 0 | 0
Pneumococcal sepsis (Infections and infestations) | 1 | 0 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Abdominal wound dehiscence (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Fibula fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Collagen disorder (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Breast cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Cholesteatoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Alcohol abuse (Psychiatric disorders) | 0 | 1 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other